CLINICAL TRIAL: NCT01794299
Title: An Exploratory, Open-label, Multicenter Study to Evaluate the Safety and Efficacy of ATIR, Donor T-lymphocytes Depleted ex Vivo of Host Alloreactive T-cells, in Patients With a Hematologic Malignancy, Who Received a CD34-selected Hematopoietic Stem Cell Transplantation From a Haploidentical Donor
Brief Title: Safety and Efficacy of Donor T-lymphocytes Depleted ex Vivo of Host Alloreactive T-cells (ATIR) in Patients With a Hematologic Malignancy Who Received a Hematopoietic Stem Cell Transplantation From a Haploidentical Donor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kiadis Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CR-AIR-007; 2012-004461-41 (EudraCT Number); File # 9427-K0980\1-21C (Other: Health Canada)
Record Dates: First submitted 2013-02-14; First posted 2013-02-18 (Estimated); Results first posted 2021-01-12 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-03

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Myelodysplastic Syndrome
Keywords: Haploidentical stem cell transplantation; Graft-versus-host disease; Immune reconstitution; Alloreactive T-cells; Photodepletion; Photodynamic treatment; TH9402; Transplant-related mortality; Hematologic malignancy
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Graft vs Host Disease; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ATIR (Experimental)
  Interventions: Biological: ATIR

INTERVENTIONS:
Biological: ATIR — Donor T-lymphocytes depleted ex vivo of host alloreactive T-cells using photodynamic treatment. Single intravenous infusion with 2x10E6 viable T-cells/kg.

SUMMARY:
The purpose of this study is to determine whether ATIR is safe and effective in reducing transplant-related mortality and improving overall survival, when infused in patients with a hematologic malignancy following a T-cell depleted stem cell graft from a related haploidentical donor.

DETAILED DESCRIPTION:
Study CR-AIR-007 is an exploratory, open-label, multicenter study. After signing informed consent, patients will receive a hematopoietic stem cell transplantation (HSCT) from a related, haploidentical donor, followed by infusion with ATIR between 28 and 32 days after the HSCT (or later if required by the patient's medical condition). Patients will receive ATIR as a single infusion at a dose of 2x10E6 viable T-cells/kg. All patients treated with ATIR will be followed up until 12 months after the HSCT. Assessments will be performed at weekly visits from the day of ATIR infusion until 8 weeks after ATIR infusion, at monthly visits from 3 until 6 months after the HSCT, every 2 months from 6 until 12 months after the HSCT, and every 6 months from 12 until 24 months after the HSCT.

ELIGIBILITY:
Inclusion Criteria:

* Any of the following hematologic malignancies: a) Acute myeloid leukemia (AML) in first remission with high-risk features or in second or higher remission b) Acute lymphoblastic leukemia (ALL) in first remission with high-risk features or in second or higher remission c) Myelodysplastic syndrome (MDS): transfusion-dependent, or intermediate or higher Revised International Prognostic Scoring System (IPSS-R) risk group
* Eligible for haploidentical stem cell transplantation according to the investigator

Exclusion Criteria:

* Availability of a suitable matched related or unrelated donor following a donor search
* In second or higher remission with the previous remission having lasted less than 6 months
* Diffusing capacity for carbon monoxide (DLCO) < 50% predicted
* Left ventricular ejection fraction < 50% (evaluated by echocardiogram or multiple gated acquisition [MUGA])
* Aspartate aminotransferase (AST) > 2.5 x upper limit of normal (ULN)(CTCAE grade 2)
* Bilirubin > 1.5 x ULN (CTCAE grade 2)
* Creatinine clearance < 50 mL/min (calculated or measured)
* Positive test for human immunodeficiency virus (HIV)
* Positive pregnancy test (women of childbearing age only)
* Prior allogeneic stem cell transplantation using stem cells from a matched sibling donor, a matched unrelated donor, a haploidentical donor, or a cord blood donor
* Prior autologous stem cell transplantation
* Stay at intensive care unit for more than 2 months in the preceding 12 months
* Estimated probability of surviving less than 3 months
* Known allergy to any of the components of ATIR (e.g., dimethyl sulfoxide)
* Any other condition which, in the opinion of the investigator, makes the patient ineligible for the study

Donor inclusion criteria

* Haploidentical family donor with 2 to 3 mismatches at the human leukocyte antigen (HLA)-A, -B and/or -DR loci of the unshared haplotype
* Male or female, age ≥ 16 and ≤ 75 years
* Eligible for donation according to the transplantation center

Donor exclusion criteria

* Positive viral test for HIV-1, HIV-2, hepatitis B virus (HBV), hepatitis C virus (HCV), Treponema pallidum, human T-lymphotropic virus (HTLV)-1*, HTLV-2*, or West Nile virus (WNV)* (if tested) (* at Canadian centers only)
* Positive pregnancy test or nursing (women of childbearing age only)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denis Claude Roy, Prof MD, Study Chair — Maisonneuve-Rosemont Hospital, Montreal Quebec
Locations (8):
- Belgium (3):
  - Algemeen Ziekenhuis Sint-Jan, Bruges
  - Université Libre de Bruxelles - Institute Jules Bordet, Brussels
  - Universitair Ziekenhuis Gasthuisberg, Leuven
- Canada (3):
  - Juravinski Hospital and Cancer Centre, Hamilton, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
- Universitätsklinikum Würzburg, Würzburg, Germany
- Hammersmith Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ATIR
Started | 31
Completed | 9
Not Completed | 22
Not completed — ATIR manufacturing not possible | 1
Not completed — Death | 14
Not completed — Graft failure | 1
Not completed — ATIR batch rejected | 2
Not completed — Relapse | 2
Not completed — Discontinued from active follow-up | 1
Not completed — Relapse and rejection of ATIR batch | 1

BASELINE CHARACTERISTICS:
Arm/Group | ATIR
Number analyzed (Participants) | 23
Age, Continuous [Median (Full Range); unit: years] | 34 [20 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Human leukocyte antigen (HLA)-match n (%) [Count of Participants; unit: Participants]
  3/6 | 16
  4/6 | 6
  5/6 | 1

OUTCOME MEASURES:

1. Primary Outcome: Transplant-related Mortality (TRM)
Description: TRM is defined as death due to causes other than disease relapse or progression, or other causes which are unrelated to the transplantation procedure (e.g. accident, suicide). The TRM rate is displayed as a function of time using the Kaplan-Meier method. The TRM rate at 6 months post HSCT is estimated from this analysis.
Time Frame: At 6 months post HSCT
Measure: Number (95% Confidence Interval); unit: Kaplan-Meier estimates (%)
Arm/Group | ATIR
Number analyzed (Participants) | 23
Kaplan-Meier estimates (%) | 13 [5 to 36]

2. Secondary Outcome: Immune Reconstitution
Description: Immunophenotyping on peripheral blood samples by means of flow cytometry assessment of immune subsets was done if the absolute lymphocyte count was higher than 0.1×10E9/l
Time Frame: Up to 24 months post HSCT
Measure: Count of Participants; unit: Participants
Arm/Group | ATIR
Number analyzed (Participants) | 23
Participants
  Number of participants with CD3 counts above 0.1×10E9/l at 24 months follow up | 18
  Number of participants with CD3 counts above 0.2×10E9/l at 24 months follow up | 13

3. Secondary Outcome: Relapse-related Mortality (RRM)
Description: Defined as death due to disease relapse or disease progression. The Kaplan-Meier analysis resulted in estimates and 95% confidence intervals (CI)s.
Time Frame: 6, 12 and 24 months post HSCT
Measure: Number (95% Confidence Interval); unit: Kaplan-Meier estimates (%)
Arm/Group | ATIR
Number analyzed (Participants) | 23
Kaplan-Meier estimates (%)
  6 months post HSCT | 5 [1 to 28]
  12 months post HSCT | 10 [3 to 35]
  24 months post HSCT | 25 [10 to 55]

4. Secondary Outcome: Overall Survival (OS)
Description: Defined as the time from HSCT until death from any cause. The Kaplan-Meier analysis resulted in estimates and 95% CIs.
Time Frame: 6, 12 and 24 months post HSCT
Measure: Number (95% Confidence Interval); unit: Kaplan-Meier estimates (%)
Arm/Group | ATIR
Number analyzed (Participants) | 23
Kaplan-Meier estimates (%)
  6 months post HSCT | 83 [60 to 93]
  12 months post HSCT | 61 [38 to 77]
  24 months post HSCT | 39 [20 to 58]

5. Secondary Outcome: Progression-free Survival (PFS)
Description: Defined as the time from HSCT until relapse, disease progression, or death, whichever occurs first. The Kaplan-Meier analysis resulted in estimates and 95% CIs.
Time Frame: 6, 12 and 24 months post HSCT
Measure: Number (95% Confidence Interval); unit: Kaplan-Meier estimates (%)
Arm/Group | ATIR
Number analyzed (Participants) | 23
Kaplan-Meier estimates (%)
  6 months post HSCT | 78 [55 to 90]
  12 months post HSCT | 61 [38 to 77]
  24 months post HSCT | 39 [20 to 58]

6. Secondary Outcome: Number of Participants With Viral, Fungal, and Bacterial Infections.
Time Frame: Up to 24 months post HSCT
Measure: Number; unit: participants
Arm/Group | ATIR
Number analyzed (Participants) | 23
participants
  Any infection, from HSCT to ATIR infusion | 17
  Any infection, from ATIR infusion to 6 months after HSCT | 19
  Any infection, from 6 months to 1 year after HSCT | 13
  Any infection, from 1 year to 2 years after HSCT | 12

7. Secondary Outcome: Number of Participants With Graft Versus Host Disease (GVHD)
Time Frame: Up to 24 months post HSCT
Measure: Number; unit: participants
Arm/Group | ATIR
Number analyzed (Participants) | 23
participants
  Any GVHD, from HSCT to ATIR infusion | 2
  Any GVHD, from ATIR infusion to 100 days after HSCT. | 0
  Any GVHD, from 100 days to 6 months after HSCT. | 3
  Any GVHD, from 6 months to 1 year after HSCT. | 3
  Any GVHD, from 1 year to 2 years after HSCT. | 4

ADVERSE EVENTS:
Arm/Group | ATIR
Serious Adverse Events (participants affected / at risk) | 3/23
Other Adverse Events (participants affected / at risk) | 4/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ATIR (N=23)
acute graft versus host disease (aGVHD) (Immune system disorders) | 1
chronic graft versus host disease (cGVHD) (Immune system disorders) | 1
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ATIR (N=23)
aGVHD (Immune system disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No